CLINICAL TRIAL: NCT03684668
Title: Psychoeducational Intervention Through Meta - Universes on Self - Efficacy in the Use of Condoms and Sexual Behavior in University Students of the Autonomous University of Chile, 2018.
Brief Title: Psychoeduc Interv. Through Meta-universes on Condom's Use Self - Efficacy and Sexual Behavior in Students of UAChile
Acronym: MVSR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection could not be completed in time and it has not been possible to continue due to the pandemic. Since it is not yet known when the face-to-face classes will resume, we moved on to the data analysis phase with the existing data.
Sponsor: Rosa Jimenez (Other)
Responsible Party: Sponsor-Investigator, Rosa Jimenez, Professor, Universidad Autónoma de Chile
Organization: Universidad Autónoma de Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SEXUALHEALTHRISKMETAVERSE
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Sexually Transmitted Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases, Bacterial
Keywords: sexual behavior; condom use; Self-Efficacy; educational technology
MeSH Terms: conditions — Sexually Transmitted Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases, Bacterial; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: This is a behavioral intervention where 120 university students will be randomly assigned to the intervention or de control group. Intervention consists in a psychoeducational activity enhanced using meta-universes or three-dimensional virtual worlds. Each selected student will undergo a three-session educational activity before a personal computer and wearing 3D lenses. The first session is called "Knowledge about STI"; the second session is entitled "Use of the male condom" and the third session is called "Talking about sexuality issues". The intervention will be carried out every 24 hours with four participants in four computers and 3D lenses available in the computer labs of the University. The control group will not receive this intervention.
Who Masked: Outcomes Assessor
Masking Description: All forms with the questionnaires will be consecutively numbered before the beginning of the study and randomly allocated to one of the study groups. This assignment list will be given to the secretary who will allocate the questionnaires to the corresponding group and deliver them to the corresponding researcher. After completion, all forms will be collected and merged and then delivered again to the secretary who will randomly assign number 1 or 2 to one of the groups and will write this number in the upper right edge of each completed questionnaire according to the original assignment list. The researcher that will introduce data in the database will include a field for this number but will not know to which of the groups it belongs. Statistical analysis will be then carried comparing groups 1 and 2. This will not be uncovered until all results are obtained and are ready for discussion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducational intervention (Experimental): The psychoeducational intervention, with the use of meta-universes,consists of three sessions in which techniques based on three of the four sources of self-efficacy described are applied.
  Interventions: Behavioral: Psychoeducational intervention
- Control (No Intervention): The control arm will not receive the psychoeducational intervention. Students in this group will complete the questionnaires before the beginning of the intervention and after its end.

INTERVENTIONS:
Behavioral: Psychoeducational intervention — The intervention will be carried out every 24 hours with four participants in four computers and 3D lenses available in the computer labs of the University.
  Arms: Psychoeducational intervention

SUMMARY:
In Chile, sexually transmitted infections (STI)s, including HIV / AIDS, are the main causes of morbidity in adolescents and young adults. The surveillance bulletin of the Institute of Public Health revealed an increase in cases of gonorrhea, over 200% in the last five years. HIV cases increased between 34% and 47% in this period as well.

Unsafe sexual behaviors are among the most important risk factors for sexually transmitted infections (STI); it has been shown that educational / behavioral interventions can achieve success in behavioral changes, especially in young people. Some studies have evaluated the effectiveness of behavioral interventions to prevent sexual risk behavior of HIV and STIs with encouraging results.

On the other hand, information and communication technologies (ICT) have been used in the prevention of STIs, HIV / AIDS. There is a considerable increase in the use of meta-universes or three-dimensional virtual worlds for educational purposes since 2006. No studies have yet been found that demonstrate the effectiveness of educational interventions carried out in meta-universes for the prevention of STIs in Chile.

This study aims to demonstrate the effectiveness of a psychoeducational intervention through the use of meta-universes, on self-efficacy in the use of condoms and safe sexual behavior, in university students.

An open randomized, controlled trial will be conducted. Dependent variables will be measured before the intervention and 15 days after the end of the intervention in the experimental group in both groups.

Students from first year to fourth year of different careers (except Nursing), currently in the Universidad Autonoma de Chile will be included after their informed consent.

The psychoeducational intervention consists of three sessions in which techniques based on three of the four sources of self-efficacy described are applied.

The intervention will be carried out every 24 hours with four participants in four computers and 3D lenses available in the computer labs of the University.

The dependent variables will be: 1) the self-efficacy in the use of male condom, measured with the Scale Condom self-efficacy scale of Brafford and Beck and 2) safe sexual behavior measured with Safe Sex Behavior Questionnaire scale of Dilorio, Lehr, Adame and Carlone. Both scales were culturally adapted to Chile.

DETAILED DESCRIPTION:
In Chile, sexually transmitted infections (STI)s, including HIV / AIDS, are the main causes of morbidity in adolescents and young adults. The surveillance bulletin of the Institute of Public Health revealed an increase in cases of gonorrhea, over 200% in the last five years. HIV cases increased between 34% and 47% in this period as well.

Unsafe sexual behaviors are among the most important risk factors for these diseases; it has been shown that educational / behavioral interventions can achieve success in behavioral changes, especially in young people. Some studies have evaluated the effectiveness of behavioral interventions to prevent sexual risk behavior of HIV and STIs with encouraging results.

On the other hand, information and communication technologies (ICT) have been used in the prevention of STIs, HIV / AIDS. These include computer interventions through meta-universes, chat rooms, text messaging and social media. There is a considerable increase in the use of meta-universes or three-dimensional virtual worlds for educational purposes since 2006. No studies have yet been found that demonstrate the effectiveness of educational interventions carried out in meta-universes for the prevention of STIs in Chile.

This study aims to demonstrate the effectiveness of a psychoeducational intervention through the use of meta-universes, on self-efficacy in the use of condoms and safe sexual behavior, in university students.

An open randomized, controlled trial will be conducted. Dependent variables will be measured before the intervention and 15 days after the end of the intervention in the experimental group, in both groups.

Students from first year to fourth year of different careers (except Nursing), currently in the Universidad Autonoma de Chile will be included after their informed consent.

The psychoeducational intervention consists of three sessions in which techniques based on three of the four sources of self-efficacy described are applied. The first session is called "Knowledge about STI"; the second session is entitled "Use of the male condom" and the third session is called "Talking about sexuality issues". In the first session screens will be created with interactive information in which the participants wearing 3D glasses will select information on different types of STIs; modeled situations will be presented in which students will perform and at the same time develop self-efficacy in terms of knowledge about STIs. In the second session four metaverses will be created, the first represents a modeled situation in which the participant selects an avatar, then selects a scenario between four risk situations where he meets a possible sexual partner. The student must select riddles that lead to responsible sexual behavior, selecting the best way to use the condom and different barrier methods, proposing its use and rejecting any risky behavior. In the third session, four meta-universes will be created through 3D technology, each participant selects an avatar and a different role is assigned to each one so that they generate sexuality communication skills among them without knowing each one's identity.

The intervention will be carried out every 24 hours with four participants in four computers and 3D lenses available in the computer labs of the University.

The dependent variables will be: 1) the self-efficacy in the use of male condom, measured with the Scale Condom self-efficacy scale of Brafford and Beck and 2) safe sexual behavior measured with Safe Sex Behavior Questionnaire scale of Dilorio, Lehr, Adame and Carlone. Both scales were culturally adapted to Chile.

ELIGIBILITY:
Inclusion Criteria:

* University students registered in the campus El Llano of the Universidad Autonoma de Chile.
* Students from first to fourth year.

Exclusion Criteria:

* Nursing students
* Medicine students

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Self-efficacy in the use of male condom | 15 days
  Self-efficacy in the use of male condom measured with an adaptation of the Condom Use Self Efficacy Scale (CUSES) developed by Brafford and Beck in 1991. This scale consists of 21 items describing an individual's feelings of confidence about being able to buy condoms, put them on and take them off, and negotiate their use with a new sexual partner. Each item is answered with a five-point Likert scale (0: total disagreement to 4: total agreement). Six items are worded negatively so should be reversed when coding. Total scores go from 0 to 84 points, the higher the better self-efficacy. This scale underwent translation and cross-cultural adaptation in Cuba (http://dx.doi.org/10.4321/S1132-12962011000200012) and is now in a process of cross-cultural validation in Chile (Universidad Autonoma de Chile) before the beginning of the study. The original authors of the scale have been consulted and agree with adaptation and validation.
Safe sexual behavior | 15 days
  Safe sexual behavior measured with an adaptation of the Safe Sex Behavior Questionnaire (SSBQ) first developed by DiIorio, Parsons, Lehr, Adame and Carlone in 1992. This scale aims to detect safe sexual practices and risky sexual behavior. The current scale has 23 items. Participants rate on a 4-point scale the degree of safe sex practices from "never" (recorded as 1) to "always" (recorded as 4). There are 8 items worded negatively that should be reversed when coding. The total possible range of scores in this adapted SSBQ is between 23 and 92, with higher scores indicating less risky sexual behavior and lower scores indicating more risky sexual behavior. This scale is undergoing translation and cross-cultural validation now in Chile (Universidad Autonoma de Chile). The original authors of the scale have been consulted and agree with adaptation and validation.

SECONDARY OUTCOMES:
Satisfaction with the intervention | one day
  Measured with a Likert scale from very unsatisfied to very satisfied (only for the intervention group)

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Hernandez, PhD, Principal Investigator — Universidad Autonoma de Chile
Locations (1):
- Universidad Autonoma de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within one year of the study completion.
Access Criteria: Data access will be released for those who request them after the publication of the study.

REFERENCES:
- [Background] Jemmott JB 3rd, Jemmott LS, O'Leary A, Ngwane Z, Icard LD, Heeren GA, Mtose X, Carty C. Cluster-randomized controlled trial of an HIV/sexually transmitted infection risk-reduction intervention for South African men. Am J Public Health. 2014 Mar;104(3):467-73. doi: 10.2105/AJPH.2013.301578. Epub 2014 Jan 16. PMID 24432923
- [Background] Khumsaen N, Stephenson R. Beliefs and Perception About HIV/AIDS, Self-Efficacy, and HIV Sexual Risk Behaviors Among Young Thai Men Who Have Sex With Men. AIDS Educ Prev. 2017 Apr;29(2):175-190. doi: 10.1521/aeap.2017.29.2.175. PMID 28467158
- [Background] Bermudez Mde L, Araujo LF, Reyes AO, Hernandez-Quero J, Teva I. Analysis of cognitive variables and sexual risk behaviors among infected and HIV-uninfected people from Spain. AIDS Care. 2016 Jul;28(7):890-7. doi: 10.1080/09540121.2016.1161163. Epub 2016 Mar 16. PMID 26981840
- [Background] Fernandez AM, Celis-Atenas K, Cordova-Rubio N, Dufey M, Correa Varella MA, Benedetti Piccoli Ferreira JH. [Youth sexuality: behaviors, attitudes and differences by sex and personality variables in Chilean university students]. Rev Med Chil. 2013 Feb;141(2):160-6. doi: 10.4067/S0034-98872013000200003. Spanish. PMID 23732487
- [Background] Gabarron E, Serrano JA, Wynn R, Armayones M. Avatars using computer/smartphone mediated communication and social networking in prevention of sexually transmitted diseases among North-Norwegian youngsters. BMC Med Inform Decis Mak. 2012 Oct 30;12:120. doi: 10.1186/1472-6947-12-120. PMID 23110684
- [Background] Ghanbarzadeh R, Ghapanchi AH, Blumenstein M, Talaei-Khoei A. A decade of research on the use of three-dimensional virtual worlds in health care: a systematic literature review. J Med Internet Res. 2014 Feb 18;16(2):e47. doi: 10.2196/jmir.3097. PMID 24550130
- [Background] Lopez LM, Otterness C, Chen M, Steiner M, Gallo MF. Behavioral interventions for improving condom use for dual protection. Cochrane Database Syst Rev. 2013 Oct 26;2013(10):CD010662. doi: 10.1002/14651858.CD010662.pub2. PMID 24163112